CLINICAL TRIAL: NCT05096338
Title: Cardiotoxicity of Prostate Cancer Therapy: Mechanisms, Predictors, and Social Determinants of Health in Prostate Cancer Patients Treated with Androgen Deprivation Therapy
Brief Title: Mechanisms, Predictors, and Social Determinants of Cardiotoxicity in Prostate Cancer
Acronym: PCT
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 12821
Record Dates: First submitted 2021-10-12; First posted 2021-10-27 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Cardiotoxicity; Drug-Related Side Effects and Adverse Reactions; Cardiovascular Diseases
Keywords: Cardiotoxicity of Chemotherapy; Cardio-Oncology; Social Determinants of Health
MeSH Terms: conditions — Prostatic Neoplasms; Cardiotoxicity; Drug-Related Side Effects and Adverse Reactions; Cardiovascular Diseases | interventions — Social Determinants of Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, and buffy coat will be banked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Social Determinants of Health — We will perform detailed phenotyping of Social Determinants of Health using the National Institute of Minority Health and Health Disparities PhenX SDOH toolkit at baseline.

SUMMARY:
This is an observational study for patients with prostate cancer that will be treated with Androgen Deprivation Therapy. The study will help the investigators learn more about how these medications affect the heart and how those effects relate to patients' medical history and social determinants of health (such as race, gender identity, education, occupation, access to health services and economic resources). Patients on this study will have echocardiograms, blood draws, and answer questions about their symptoms and activity level. Patients will be followed on this study for up to 5 years.

DETAILED DESCRIPTION:
The investigators propose a prospective longitudinal cohort of prostate cancer patients treated with Androgen Deprivation Therapy (ADT) to determine the associations between social determinants of health (SDOH) and cardiotoxicity risk and to determine wither associations between SDOH and cardiotoxicity risk differs according to race. Patients will be followed with serial echo, blood draw, and surveys prior to start of ADT and then 6 months, 1 year, 2 years, 3 years, and 5 years after start of ADT.

ELIGIBILITY:
Inclusion Criteria:

Men older than 18 years of age Prostate cancer diagnosis planned for treatment with ≥6 months of ADT (with or without RT) for clinically localized, biochemically recurrent, or oligometastatic disease. Planned ADT regimens may include: GnRH agonists (goserelin, histrelin, leuprolide, triptorelin) with or without first-generation anti-androgens and GnRH antagonists (degarelix). Additional systemic agents, including second-generation androgen receptor signaling inhibitors, may be used in combination with GnRH agonist/antagonist therapies per provider clinical discretion.

Ability to provide informed consent

Exclusion Criteria:

Prior ADT injection within 6 months prior to enrollment Inability or unwillingness to provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the medical oncology practices at the Abramson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | through study completion (expected to be 15 years)
  Absolute change in LVEF by echocardiogram at follow-up

SECONDARY OUTCOMES:
Cancer therapy-related cardiac dysfunction (CTRCD) | through study completion (expected to be 15 years)
  Incidence of CTRCD defined as at least a 10% absolute change in LVEF by echocardiogram at follow-up relative to baseline to a value < 50%
Symptomatic Heart Failure (HF) | through study completion (expected to be 15 years)
  Incidence of symptomatic heart failure (centrally adjudicated)
Change in Longitudinal Strain | through study completion (expected to be 15 years)
  Change in longitudinal strain by echo from baseline
Change in Circumferential Strain | through study completion (expected to be 15 years)
  Change in circumferential strain by echo from baseline
Change in Diastolic function | through study completion (expected to be 15 years)
  Change in diastolic function defined as E/e' by echo from baseline
Change in Left Ventricular (LV) Mass | through study completion (expected to be 15 years)
  Change in LV Mass by echo from baseline
Change in Relative LV Wall Thickness | through study completion (expected to be 15 years)
  Change in relative LV wall thickness from baseline
Change in Ventricular-Arterial Coupling | through study completion (expected to be 15 years)
  Change in Ventricular-Arterial Coupling defined as Ea/Ees by echo from baseline
Change in LV Twist | through study completion (expected to be 15 years)
  Change in LV Twist measured by 3D echo from baseline
Change in LV Torsion | through study completion (expected to be 15 years)
  Change in LV Torsion measured by 3D echo from baseline
Change in NTproBNP | through study completion (expected to be 15 years)
  Change in NTproBNP measured in batches from banked samples from baseline.
Change in high-sensitivity troponin (hsTnT) | through study completion (expected to be 15 years)
  Change in hs-TnT measured in batches from banked samples from baseline.
Change in patient reported fatigue | through study completion (expected to be 15 years)
  Change in Patient Reported Outcomes Information System (PROMIS) Fatigue Score from baseline. A higher score corresponds to higher reported levels of fatigue.
Change in patient reported quality of life | through study completion (expected to be 15 years)
  Change in Patient Reported Outcomes Information System (PROMIS) Global Health score from baseline. Higher scores indicate a healthier patient.
Change in patient reported activity level | through study completion (expected to be 15 years)
  Change in total weekly leisure activity in METS assessed by Godin Leisure Time Exercise Questionnaire from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barrett M, Wilcox NS, Huang A, Levy R, Demissei B, Narayan V, Ky B. Bearing allostatic load: insights into a more equitable future within cardio-oncology. Trends Mol Med. 2022 Dec;28(12):1040-1049. doi: 10.1016/j.molmed.2022.09.006. Epub 2022 Oct 4. PMID 36207229